CLINICAL TRIAL: NCT02957214
Title: Prospective Controlled Study of the Effects of an Intervention Program Based on Pain Education in Pain Activity Patterns and Brain Connectivity in Patients With Chronic Pelvic Pain by Magnetic Resonance Images
Brief Title: Effects of an Intervention Program Based on Pain Education in Patients With Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rafael Torres Cueco, PT, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-27072016
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain education (Experimental): The patient education provides a basic set of information that includes the explanation of possible pathophysiological mechanisms involved in the development of chronic pain. The main objective is to reduce pain threatening and alarmist interpretation. The patient must understand that the pain is not necessarily a sign of injury, but the consequence of a maladaptive central sensitization. One element of this therapeutic strategy is to help the patient to perform physical activities that involve a gradual exposition to stimuli associated with their pain and promote physical recovery exposure. Pain education also aims to reduce fear-avoidance behavior and the patient's disability.
  Interventions: Other: Pain education

INTERVENTIONS:
Other: Pain education — The patient education provides a basic set of information that includes the explanation of possible pathophysiological mechanisms involved in the development of chronic pain. The main objective is to reduce pain threatening and alarmist interpretation. The patient must understand that the pain is not necessarily a sign of injury, but the consequence of a maladaptive central sensitization. One element of this therapeutic strategy is to help the patient to perform physical activities that involve a gradual exposition to stimuli associated with their pain and promote physical recovery exposure. Pain education also aims to reduce fear-avoidance behavior and the patient's disability.
  Other Names: pain neuroscience education

SUMMARY:
The purpose of this study is to obtain imaging biomarkers based on changes in activity patterns and changes in brain connectivity obtained with the analysis of functional magnetic resonance imaging (fMRI) and tractography that are related to chronic pelvic pain

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Chronic pelvic pain diagnosis
* Pain duration > 6 months
* Average pain intensity ≥ 6 during the previous week

Exclusion Criteria:

* Suspected or knowledge of actual organic pathology that requires medical or surgical treatment
* Psychiatric illness: major depression, bipolar syndrome...
* Patients with significant cognitive deficits
* Have pacemaker, metal prostheses or hearing aids incompatible with MRI
* Severe traumatic brain injury
* Previous cranial surgeries
* History of alcoholism
* Do not sign informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Study Functional Magnetic Resonance Image (fMRI) | At day 1
  Fractional anisotropy maps Functional MRI Voxel voxel orientation maps Maps diffusivity Functional study RestingState
Study Functional Magnetic Resonance Image (fMRI) | Between 7 and 31 days later randomly
  Fractional anisotropy maps Functional MRI
Study Functional Magnetic Resonance Image (fMRI) | At 6 months of completing the education program
  Fractional anisotropy maps Functional MRI

SECONDARY OUTCOMES:
numerical rating scale NRS | Day 1 and at 6 months of completing the education program
Multidimensional Pain Inventory (MPI) - Interference Scale | Day 1 and at 6 months of completing the education program
Oswestry Disability Index (ODI) | Day 1 and at 6 months of completing the education program
Hospital Anxiety and Depression Scale (HADS) | Day 1 and at 6 months of completing the education program
Pain Catastrophizing Scale | Day 1 and at 6 months of completing the education program
Tampa Scale for Kinesiophobia-11 | Day 1 and at 6 months of completing the education program
Female Sexual Function Index | Day 1 and at 6 months of completing the education program

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Torres-Cueco, Principal Investigator
Locations (1):
- Rafael Torres Cueco, Valencia, Spain